CLINICAL TRIAL: NCT01884545
Title: Genetic Risk and Health Coaching for Type 2 Diabetes and Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00039569
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2017-03

CONDITIONS: Coronary Heart Disease, Susceptibility to, 5; Prediabetic State
Keywords: heart disease; type 2 diabetes; genetic testing; health coaching; risk assessment
MeSH Terms: conditions — Coronary Disease; Prediabetic State; Heart Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (4):
- Standard Risk Assessment (SRA) (Active Comparator): Subjects will receive a standard risk assessment only for coronary heart disease (CHD) and type 2 diabetes (T2D). Standard risk factors are reviewed by a provider at a risk counseling visit with the subject.
  Interventions: Behavioral: Standard risk assessment
- SRA plus Health Coaching (HC) (Experimental): In addition to the standard risk assessment for CHD and T2D subjects will receive health coaching intervention for 6 months
  Interventions: Behavioral: Health coaching; Behavioral: Standard risk assessment
- SRA plus Genetic Risk Counseling (GRC) (Experimental): In addition to the SRA subjects will receive genetic risk counseling at the risk counseling visit with a clinic provider. Genetic test results for CHD (rs10757274) and T2D (rs7903146, rs1801282, rs5219) risk variants will be incorporated into the risk profile reviewed with subjects.
  Interventions: Genetic: Genetic risk counseling; Behavioral: Standard risk assessment
- SRA+HC+GRC (Experimental): In addition to the standard risk assessment for CHD and T2D subjects will receive genetic risk counseling and health coaching intervention for 6 months.
  Interventions: Behavioral: Health coaching; Genetic: Genetic risk counseling; Behavioral: Standard risk assessment

INTERVENTIONS:
Behavioral: Health coaching — Telephonic health coaching sessions with a trained certified health coach for a period of 6 months (total of 10 biweekly calls).
  Arms: SRA plus Health Coaching (HC); SRA+HC+GRC
Genetic: Genetic risk counseling — In addition to the SRA subjects will receive genetic risk counseling at the risk counseling visit with a clinic provider. Genetic test results for CHD (rs10757274) and T2D (rs7903146, rs1801282, rs5219) risk variants will be incorporated into the risk profile reviewed with subjects.
  Arms: SRA plus Genetic Risk Counseling (GRC); SRA+HC+GRC
Behavioral: Standard risk assessment — Standard risk assessment for coronary heart disease (CHD) and type 2 diabetes (T2D). Standard risk factors are reviewed by a provider at a risk counseling visit with the subject.

SUMMARY:
The purpose of this study is to examine whether the use of genetic test information and/or health coaching in patient risk counseling for heart disease and diabetes affect health behaviors and health outcomes in active-duty Air Force (ADAF), beneficiaries or dependents and Air Force retiree patients.

Total of 400 subjects will be enrolled. They will be randomly(like flipping a coin)assigned to 4 groups: 1)Standard risk assessment (SRA)only; 2)SRA plus genetic risk information (SRA+G); 3)SRA plus health coaching (SRA+HC); or 4)SRA, genetic risk information, and health coaching (SRA+G+HC). Subjects randomized to the two genetic arms will have blood collected for testing of investigational coronary heart disease (CHD) and type 2 diabetes (T2D) risk markers. Participants in the two groups that include health coaching will be assigned to a trained certified health coach for a period of 6 months. The duration of the study is 12 months with 3 in person visits (baseline, 6 months and 12 months) and completion of surveys at 6 weeks and 3 month time points.

DETAILED DESCRIPTION:
This study will examine the impact of providing genetic CHD and T2D risk information, with or without a supportive behavioral intervention, on promoting risk-reducing behaviors and improving clinical outcomes. In short, using a 4-group (2X2) randomized controlled trial (RCT) design, this study will determine whether incorporating multiple-marker genetic testing into risk counseling for CHD and T2D, coupled with a health coaching intervention will lead to greater changes in physical fitness, health behaviors, risk status and clinical outcomes in active-duty Air Force (ADAF), beneficiaries or dependents and AF retiree patients (N=400).

The study will address the following task objectives:

1. Determine the main and interactive effects of multiple-marker genetic risk information incorporated into standard CHD and T2D risk counseling (Standard Risk Assessment, or SRA) and an established, structured telephonic health coaching intervention on health behavior change (diet, exercise habits, smoking cessation) over 12 months, with a focus on ADAF patients, as well as their beneficiaries and retirees.
2. Determine the main and interactive effects of genetic risk information incorporated into standard CHD and T2D risk counseling and a telephonic health coaching intervention on clinical outcomes (fasting blood glucose, blood pressure, BMI, LDL, triglycerides, total cholesterol, AF composite fitness scores) over 12 months in this AF cohort.

   Given the lack of RCTs on the effects of differing genetic test results, such as false reassurance and genetic determinism, we will also pursue a third, exploratory task objective:
3. Examine the differential effects of level of CHD and T2D genetic risk (# of risk alleles) on behavior change (diet, exercise habits, smoking cessation) and AF fitness scores at 12 months post baseline.

Baseline data collection: After screening and informed consent, height and weight, SBP, waist circumference, current lab results (FPG, total cholesterol, triglycerides, LDL, HbA1c, and HDL) and current PHA (physical health assessment) data with fitness scores ( for active duty personnel only) will be obtained from the medical records. Subjects randomized to the two genetic arms will have blood collected for testing of investigational CHD and T2D risk markers.

Randomization will take place to one of the following: SRA only; SRA plus genetic risk information (SRA+G); SRA plus health coaching (SRA+HC); or SRA, genetic risk information, and health coaching (SRA+G+HC).

Risk Counseling Visit: Within four weeks after the baseline visit all participants will receive risk counseling with trained provider(s) at each clinic site.

Health coaching intervention: Participants in the two groups that include health coaching will be assigned to a trained health coach for a period of 6 months (n=200). IHC (Integrative Health Coaching) sessions will be provided by telephone using a structure that has evolved in multiple trials and clinical programs at Duke Integrative Medicine.

Six week, 3-, and 6-month follow-ups: At 6 weeks, 3 months and 6 months after the baseline visit, participants will be asked to complete selected surveys online.

6month and 12 month study visits: 12 months from the baseline visit, active duty participants will complete their annual PHA, required annual AF fitness testing; and all participants will complete study visits at 6 and 12 months for weight, waist circumference, BP, fasting glucose or HbA1c and lipid panels to be re-assessed. Surveys will be completed at or prior to the final 12 month visit as well.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Willingness and ability to provide informed consent
* Have an active email address and internet access
* Physical exam in the last 12 months with the following documented evaluations in EMR (Electronic Medical record):

  1. Blood pressure
  2. Height and weight
  3. Fasting blood glucose or Hemoglobin A1C (HbA1c)
  4. Lipid panel (TC, LDL, HDL, TRIG) with at least one of them outside of the normal ranges defined as:

  i.BMI ≥ 25 kg/m2 (BMI = weight [kg] / ht [m]2)

ii.FPG > 100 AND ≤ 125 mg/dL

iii.HbA1c > 5.7% ≤ 6.4%

iv.SBP ≥ 130 mmHg

v.TC ≥ 200 mg/dL

vi.TRIG ≥ 150 mg/dL

vii.LDL ≥ 129 mg/dL

Exclusion Criteria:

* Projected deployment in the upcoming 6 months
* Diagnosed type 2 diabetes
* Diagnosed coronary heart disease (CHD) -(Myocardial Infarction, or documented CHD)
* Inability to ambulate or participate in physical activity
* Serious chronic disease related complications or conditions that could significantly affect study outcomes [currently treated cancer, renal failure, cardiovascular accident (CVA) with residual effects on functioning
* Current participation in another research study
* Spouse, partner or other household member already participating in this study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-07; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Vorderstrasse, DNSc, Principal Investigator — Duke University, School of Nursing; Ruth Wolever, PhD, Principal Investigator — Duke University, Duke Intergrative Medicina
Locations (1):
- David Grant Medical Center, Fairfield, California, United States

REFERENCES:
- [Background] Palomaki GE, Melillo S, Bradley LA. Association between 9p21 genomic markers and heart disease: a meta-analysis. JAMA. 2010 Feb 17;303(7):648-56. doi: 10.1001/jama.2010.118. PMID 20159873
- [Background] McCarthy MI. Genomics, type 2 diabetes, and obesity. N Engl J Med. 2010 Dec 9;363(24):2339-50. doi: 10.1056/NEJMra0906948. No abstract available. PMID 21142536
- [Background] Florez JC, Jablonski KA, Bayley N, Pollin TI, de Bakker PI, Shuldiner AR, Knowler WC, Nathan DM, Altshuler D; Diabetes Prevention Program Research Group. TCF7L2 polymorphisms and progression to diabetes in the Diabetes Prevention Program. N Engl J Med. 2006 Jul 20;355(3):241-50. doi: 10.1056/NEJMoa062418. PMID 16855264
- [Background] Sheridan SL, Viera AJ, Krantz MJ, Ice CL, Steinman LE, Peters KE, Kopin LA, Lungelow D; Cardiovascular Health Intervention Research and Translation Network Work Group on Global Coronary Heart Disease Risk. The effect of giving global coronary risk information to adults: a systematic review. Arch Intern Med. 2010 Feb 8;170(3):230-9. doi: 10.1001/archinternmed.2009.516. PMID 20142567
- [Background] Brautbar A, Ballantyne CM, Lawson K, Nambi V, Chambless L, Folsom AR, Willerson JT, Boerwinkle E. Impact of adding a single allele in the 9p21 locus to traditional risk factors on reclassification of coronary heart disease risk and implications for lipid-modifying therapy in the Atherosclerosis Risk in Communities study. Circ Cardiovasc Genet. 2009 Jun;2(3):279-85. doi: 10.1161/CIRCGENETICS.108.817338. Epub 2009 Apr 21. PMID 20031596
- [Result] Vorderstrasse AA, Ginsburg GS, Kraus WE, Maldonado MC, Wolever RQ. Health coaching and genomics-potential avenues to elicit behavior change in those at risk for chronic disease: protocol for personalized medicine effectiveness study in air force primary care. Glob Adv Health Med. 2013 May;2(3):26-38. doi: 10.7453/gahmj.2013.035. PMID 24416670
- [Derived] Lee C, Yang Q, Vorderstrasse A, Wolever RQ. Health Coaching Impacts Stage-Specific Transitions in Multiple Health Behaviors for Patients at High Risk for Coronary Heart Disease and Type 2 Diabetes: A Multigroup Latent Transition Analysis. J Cardiovasc Nurs. 2025 Sep-Oct 01;40(5):E220-E230. doi: 10.1097/JCN.0000000000001154. Epub 2024 Oct 24. PMID 39454076
- [Derived] Lee C, Wolever RQ, Min SH, Vorderstrasse AA, Yang Q. Network Psychometrics of the 10-Item Perceived Stress Scale Among Patients With High Cardiovascular and Type 2 Diabetes Risk Using Exploratory Graph Analysis. J Cardiovasc Nurs. 2024 Mar-Apr 01;39(2):E36-E43. doi: 10.1097/JCN.0000000000000996. Epub 2023 May 29. Dutch, English. PMID 37249540
- [Derived] Yang Q, Zhao A, Lee C, Wang X, Vorderstrasse A, Wolever RQ. Latent Profile/Class Analysis Identifying Differentiated Intervention Effects. Nurs Res. 2022 Sep-Oct 01;71(5):394-403. doi: 10.1097/NNR.0000000000000597. Epub 2022 Apr 14. PMID 35417442

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 220 subjects were consented. Prior to randomization 9 subjects withdrew from the study, 10 were lost to follow up, and 1 did not meet inclusion criteria. 200 participants were randomized.
Period: Overall Study
Arm/Group | Standard Risk Assessment (SRA) | SRA Plus Health Coaching (HC) | SRA Plus Genetic Risk Counseling (GRC) | SRA+HC+GRC
Started | 50 | 49 | 49 | 52
Completed | 37 | 31 | 35 | 43
Not Completed | 13 | 18 | 14 | 9
Not completed — Lost to Follow-up | 6 | 4 | 9 | 4
Not completed — Patient withdrawn | 7 | 12 | 5 | 5
Not completed — Non-adherence | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Risk Assessment (SRA) | SRA Plus Health Coaching (HC) | SRA Plus Genetic Risk Counseling (GRC) | SRA+HC+GRC | Total
Number analyzed (Participants) | 50 | 49 | 49 | 52 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.16 (10.92) | 48.67 (12.67) | 48.35 (10.51) | 44.85 (11.85) | 47.72 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 31 | 20 | 98
  Male | 28 | 24 | 18 | 32 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 2 | 5 | 18
  Not Hispanic or Latino | 40 | 45 | 47 | 47 | 179
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 9 | 12 | 13 | 5 | 39
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2 | 0 | 4
  Black or African American | 8 | 8 | 7 | 6 | 29
  White | 29 | 29 | 25 | 36 | 119
  More than one race | 1 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 49 | 49 | 52 | 200
Dietary Intake (Percent energy from fat) [Mean (Standard Deviation); unit: percent] | 34.50 (3.60) | 34.87 (3.17) | 34.13 (4.55) | 35.66 (4.91) | 34.81 (4.14)
Dietary Intake (Daily grams of fiber) [Mean (Standard Deviation); unit: grams] | 16.65 (5.82) | 14.94 (5.57) | 15.75 (5.83) | 18.27 (8.68) | 16.46 (6.73)
Physical Activity [Count of Participants; unit: Participants]
  Inactive/light intensity activity | 26 | 20 | 25 | 25 | 96
  Moderate/ hard/very hard intensity activity | 24 | 29 | 24 | 27 | 104
Smoking Status [Count of Participants; unit: Participants]
  No | 45 | 46 | 44 | 43 | 178
  Yes | 5 | 3 | 5 | 9 | 22
Medication Adherence (Morisky 4) [Count of Participants; unit: Participants] — The Medication Adherence (Morisky 4) data was only collected for patients who were taking medication
  Participants
    Low Adherence | 16 | 12 | 19 | 14 | 61
    Medium Adherence | 13 | 12 | 12 | 15 | 52
    High Adherence | 13 | 17 | 11 | 15 | 56
    Not applicable (patient not taking medication) | 8 | 7 | 7 | 8 | 30
Weight [Mean (Standard Deviation); unit: kg] | 85.94 (17.05) | 82.15 (16.75) | 84.96 (20.66) | 89.07 (17.76) | 85.58 (18.15)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 98.86 (10.73) | 98.51 (16.42) | 97.23 (13.50) | 98.56 (12.09) | 98.30 (13.23)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 128.60 (11.06) | 126.41 (13.03) | 123.24 (10.87) | 128.68 (13.30) | 126.77 (12.24)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 80.78 (8.89) | 80.77 (10.38) | 78.26 (8.36) | 80.62 (10.70) | 80.12 (9.63)
High-density Lipoprotein (HDL) [Mean (Standard Deviation); unit: mg/dL] | 53.66 (17.15) | 56.45 (18.62) | 49.59 (13.50) | 50.50 (16.41) | 52.53 (16.62)
Low-density Lipoprotein (LDL) [Mean (Standard Deviation); unit: mg/dL] | 133.63 (32.05) | 133.51 (42.40) | 131.94 (32.90) | 136.95 (37.15) | 134.05 (36.12)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 176.19 (123.80) | 150.73 (70.53) | 157.35 (87.76) | 156.60 (69.44) | 160.24 (90.33)

OUTCOME MEASURES:

1. Primary Outcome: Dietary Intake as Measured by Percent Energy From Fat
Description: Dietary intake as measured by percent energy from fat, adjusted for baseline
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: percent energy from fat
Groups:
- Health Coaching: Participants who received health coaching
- Non-Health Coaching: Participants who did not receive health coaching
- Genetic Risk Counseling: Patients who received genetic risk counseling
- Non-Genetic Risk Counseling: Patients who did not receive genetic risk counseling
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
percent energy from fat | 33.75 (0.5) | 34.9 (0.5) | 33.72 (0.47) | 35.05 (0.52)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.1073, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.0615, Regression, Linear

2. Primary Outcome: Dietary Intake as Measured by Daily Grams of Fiber
Description: Dietary intake as measured by daily grams of fiber, adjusted for baseline
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
grams | 15.69 (0.51) | 15.38 (0.51) | 15.24 (0.49) | 15.89 (0.54)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.6732, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.3754, Regression, Linear

3. Primary Outcome: Physical Activity, as Measured by the Stanford Brief Activity Survey (SBAS)
Description: The Stanford Brief Activity Survey is a 2-item survey that assesses two categories of physical activity - work and leisure. There are five options for degree of activity to choose from in each of the two areas of activity. Activity categories (inactive, light-intensity activity, moderate-intensity activity, hard-intensity activity, and very hard-intensity) are represented in a table of different patterns. Degree of work activity is represented on the vertical axis and degree of leisure activity is represented on the horizontal axis. The overall activity level category is determined by where the two responses intersect.
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol. Some participants were not analyzed because data were missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 72 | 72 | 77 | 67
Participants
  Inative/light intensity activity | 25 | 41 | 34 | 32
  moderate intensity activity | 30 | 18 | 23 | 25
  hard/very hard intensity activity | 17 | 13 | 20 | 10
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.0073, Regression, Logistic; Odds Ratio (OR) = 2.853, 95% CI 2-sided [1.326 to 6.139]
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.9068, Regression, Logistic; Odds Ratio (OR) = 1.045, 95% CI 2-sided [0.5 to 2.183]

4. Primary Outcome: Smoking Status
Time Frame: 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 69 | 66 | 71 | 64
Participants
  Smoked in the last 30 days = No | 65 | 63 | 67 | 61
  Smoked in the last 30 days = Yes | 4 | 3 | 4 | 3
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.7822, Regression, Logistic; Odds Ratio (OR) = 1.333, 95% CI 2-sided [0.173 to 10.254]
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.7822, Regression, Logistic; Odds Ratio (OR) = 1.333, 95% CI 2-sided [0.173 to 10.254]

5. Primary Outcome: Medication Adherence as Measured by Morisky Adherence Survey MMAS8
Description: Scores of the MMAS-8 range from 0 to 8. A score below 6 indicates low adherence, a score between 6 < 8 medium adherence and a score of 8 high adherence.
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
units on a scale | 6.66 (0.19) | 6.59 (0.18) | 6.79 (0.17) | 6.43 (0.19)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.7985, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.1642, Regression, Linear

6. Primary Outcome: Weight
Description: Weight in kg
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
kg | 86.61 (0.43) | 86.76 (0.45) | 86.77 (0.43) | 86.59 (0.45)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.8027, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.7751, Regression, Linear

7. Primary Outcome: Waist Circumference
Description: Waist circumference in cm
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
cm | 97.43 (0.63) | 96.9 (0.64) | 97.29 (0.62) | 97.04 (0.65)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.5557, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.7834, Regression, Linear

8. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure in mmHg
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
mmHg | 124.47 (1.21) | 127.05 (1.25) | 124.71 (1.2) | 126.83 (1.26)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.1439, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.2275, Regression, Linear

9. Primary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure in mmHg
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
mmHg | 79.79 (0.95) | 79.38 (0.98) | 79.59 (0.95) | 79.59 (0.99)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.7639, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.9999, Regression, Linear

10. Primary Outcome: High-density Lipoprotein (HDL)
Description: High-density lipoprotein (HDL) in mg/dL
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
mg/dL | 54.27 (0.93) | 53.3 (0.96) | 53.02 (0.93) | 54.67 (0.99)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.4673, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.2297, Regression, Linear

11. Primary Outcome: Low-density Lipoprotein (LDL)
Description: Low-density lipoprotein (LDL) in mg/dL
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
mg/dL | 128.62 (3.5) | 122.42 (3.6) | 125.33 (3.47) | 125.93 (3.68)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.2192, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.9062, Regression, Linear

12. Primary Outcome: Triglycerides
Description: Triglycerides in mg/dL
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
mg/dL | 149.34 (6.67) | 135.36 (6.87) | 148.3 (6.59) | 136.09 (7)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.1466, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.2070, Regression, Linear

13. Secondary Outcome: Fasting Blood Glucose
Description: Adjusted for baseline
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
mg/dL | 99.62 (1.54) | 100.64 (1.42) | 100.13 (1.44) | 100.23 (1.56)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.6289, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.9631, Regression, Linear

14. Secondary Outcome: Body Mass Index (BMI)
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
kg/m2 | 28.97 (0.25) | 29.4 (0.25) | 29.22 (0.25) | 29.14 (0.26)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.2313, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.8029, Regression, Linear

15. Secondary Outcome: Total Cholesterol
Description: Adjusted for baseline
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
mg/dL | 212.86 (4.01) | 202.39 (4.1) | 207.07 (3.99) | 208.51 (4.27)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.0710, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.8069, Regression, Linear

16. Secondary Outcome: AF Composite Fitness Scores
Description: Last annual fitness exam result, collected as pass or fail
Time Frame: 12 months
Population: Data only collected on active duty participants as part of their annual assessment. Randomization Arms/Groups were regrouped as pre-specified in the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 22 | 6 | 18 | 10
Participants
  Fail | 0 | 1 | 1 | 0
  Pass | 22 | 5 | 17 | 10
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.0512, Chi-squared
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.4478, Chi-squared

17. Secondary Outcome: Framingham Risk Score (FRS)
Time Frame: 12 months
Population: risk score data was only collected and calculated at baseline
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Diabetes Risk Score
Time Frame: 12 months
Population: risk score data was only collected and calculated at baseline
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Secondary Outcome: Perceived Risk for Coronary Heart Disease (CHD)
Description: Investigator developed questions assessing level of personal perceived risk, fear, anger, worry regarding CHD risk. The consequences subscale ranges from 6-30. Higher scores on the consequences represent strongly held beliefs about negative consequences of the illness. The personal control subscale ranges from 6-30 and the treatment control subscale ranges from 2-10. Higher scores on the personal control and treatment control represent positive beliefs about the controllability of the illness. The emotional representations scores range from 6-30. Higher score indicates higher levels of worry or anxiety about risk of illness.
Time Frame: 6 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
units on a scale
  Consequences subscale | 23.35 (0.53) | 23.55 (0.53) | 24.03 (0.52) | 22.83 (0.53)
  Personal control | 25.44 (0.38) | 24.42 (0.39) | 25.15 (0.38) | 24.62 (0.39)
  Treatment control | 8.44 (0.13) | 8.21 (0.13) | 8.39 (0.12) | 8.23 (0.13)
  Emotional representations | 13.54 (0.37) | 14.15 (0.37) | 13.68 (0.36) | 14 (0.37)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Perceived Risk for CHD, Consequences subscale; Test type: Superiority; p = 0.7923, Regression, Linear
Statistical Analysis 2: Comparison: Health Coaching vs Non-Health Coaching; Perceived Risk for CHD, Personal control; Test type: Superiority; p = 0.0636, Regression, Linear
Statistical Analysis 3: Comparison: Health Coaching vs Non-Health Coaching; Perceived Risk for CHD, Treatment control; Test type: Superiority; p = 0.2063, Regression, Linear
Statistical Analysis 4: Comparison: Health Coaching vs Non-Health Coaching; Perceived Risk for CHD, Emotional representations; Test type: Superiority; p = 0.2529, Regression, Linear
Statistical Analysis 5: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Perceived Risk for coronary heart disease (CHD), Consequences subscale; Test type: Superiority; p = 0.1085, Regression, Linear
Statistical Analysis 6: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Perceived Risk for coronary heart disease (CHD), personal control subscale; Test type: Superiority; p = 0.3370, Regression, Linear
Statistical Analysis 7: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Perceived Risk for coronary heart disease (CHD), treatment control subscale; Test type: Superiority; p = 0.3483, Regression, Linear
Statistical Analysis 8: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Perceived Risk for coronary heart disease (CHD), emotional representations; Test type: Superiority; p = 0.5384, Regression, Linear

20. Secondary Outcome: Perceived Risk for Type 2 Diabetes (T2D)
Description: Investigator developed questions assessing level of personal perceived risk, fear, anger, worry regarding T2D risk. The consequences subscale ranges from 6-30. Higher scores on the consequences represent strongly held beliefs about negative consequences of the illness. The personal control subscale ranges from 6-30 and the treatment control subscale ranges from 2-10. Higher scores on the personal control and treatment control represent positive beliefs about the controllability of the illness. The emotional representations scores range from 6-30. Higher score indicates higher levels of worry or anxiety about risk of illness.
Time Frame: 6 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
units on a scale
  Consequences subscale | 22.05 (0.55) | 21.79 (0.56) | 22.32 (0.54) | 21.63 (0.56)
  Personal control | 24.79 (0.36) | 24.55 (0.36) | 25.14 (0.35) | 24.28 (0.36)
  Treatment control | 8.37 (0.14) | 8.18 (0.14) | 8.35 (0.13) | 8.2 (0.14)
  Emotional representations | 13.23 (0.36) | 14.66 (0.37) | 13.75 (0.37) | 14.18 (0.37)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Perceived Risk for T2D, Consequences subscale; Test type: Superiority; p = 0.7447, Regression, Linear
Statistical Analysis 2: Comparison: Health Coaching vs Non-Health Coaching; Perceived Risk for T2D, Personal control; Test type: Superiority; p = 0.6378, Regression, Linear
Statistical Analysis 3: Comparison: Health Coaching vs Non-Health Coaching; Perceived Risk for T2D, Treatment control; Test type: Superiority; p = 0.3209, Regression, Linear
Statistical Analysis 4: Comparison: Health Coaching vs Non-Health Coaching; Perceived Risk for T2D, Emotional representations; Test type: Superiority; p = 0.0058, Regression, Linear
Statistical Analysis 5: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Perceived Risk for type 2 diabetes (T2D), Consequences subscale; Test type: Superiority; p = 0.3769, Regression, Linear
Statistical Analysis 6: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Perceived Risk for type 2 diabetes (T2D), personal control; Test type: Superiority; p = 0.0872, Regression, Linear
Statistical Analysis 7: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Perceived Risk for type 2 diabetes (T2D), treatment control; Test type: Superiority; p = 0.4302, Regression, Linear
Statistical Analysis 8: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Perceived Risk for type 2 diabetes (T2D), emotional representations; Test type: Superiority; p = 0.4133, Regression, Linear

21. Secondary Outcome: Patient Activation Score
Description: Patient activation is the degree to which patients accept an active role in their healthcare, and have the knowledge, skills and confidence to take care of their health. When scored as a continuous variable, the range is from 0 to 100, with higher numbers indicating greater levels of patient activation.
Time Frame: 12 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
units on a scale | 73.13 (1.5) | 70.95 (1.53) | 72.3 (1.45) | 71.51 (1.55)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.3106, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.7087, Regression, Linear

22. Secondary Outcome: Stages of Change
Description: These evidence-based questions are validated and based upon the Transtheoretical Model and assess an individual's readiness to make behavioral change in 5 health behavior domains (dietary intake, exercise, weight loss, smoking cessation, and medication adherence).
Time Frame: 6 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
Participants
  Weight reduction: Pre-contemplation | 2 | 1 | 1 | 2
  Weight reduction: Contemplation | 8 | 10 | 8 | 10
  Weight reduction: Preparation | 4 | 3 | 4 | 3
  Weight reduction: Action | 47 | 43 | 53 | 37
  Weight reduction: Maintenance | 10 | 11 | 8 | 13
  Exercise behavior: Pre-contemplation | 2 | 3 | 1 | 4
  Exercise behavior: Contemplation | 9 | 16 | 10 | 15
  Exercise Behavior: Preparation | 15 | 20 | 18 | 17
  Exercise Behavior: Action | 29 | 23 | 26 | 26
  Exercise Behavior: Maintenance | 20 | 13 | 21 | 12
  Smoking behavior: Pre-contemplation | 2 | 1 | 1 | 2
  Smoking behavior: Contemplation | 2 | 2 | 3 | 1
  Smoking behavior: Preparation | 3 | 2 | 4 | 1
  Smoking behavior: Action | 4 | 5 | 5 | 4
  Healthier eating behavior: Pre-contemplation | 2 | 0 | 1 | 1
  Healthier eating behavior: Contemplation | 8 | 9 | 9 | 8
  Healthier eating behavior: Preparation | 6 | 7 | 8 | 5
  Healthier eating behavior: Action | 41 | 44 | 41 | 44
  Healthier eating behavior: Maintenance | 13 | 11 | 13 | 11
  Stress behavior: Pre-contemplation | 7 | 4 | 4 | 7
  Stress behavior: Contemplation | 9 | 10 | 9 | 10
  Stress behavior: Preparation | 8 | 4 | 8 | 4
  Stress behavior: Action | 27 | 23 | 22 | 28
  Stress behavior: Maintenance | 24 | 34 | 33 | 25
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Stages of Change, Weight reduction; Test type: Superiority; p = 0.9259, Regression, Logistic; Odds Ratio (OR) = 1.034, 95% CI 2-sided [0.511 to 2.094]
Statistical Analysis 2: Comparison: Health Coaching vs Non-Health Coaching; Stages of Change, Exercise behavior; Test type: Superiority; p = 0.0082, Regression, Logistic; Odds Ratio (OR) = 2.252, 95% CI 2-sided [1.234 to 4.111]
Statistical Analysis 3: Comparison: Health Coaching vs Non-Health Coaching; Stages of Change, Smoking behavior; Test type: Superiority; p = 0.2954, Regression, Logistic; Odds Ratio (OR) = 0.423, 95% CI 2-sided [0.084 to 2.120]
Statistical Analysis 4: Comparison: Health Coaching vs Non-Health Coaching; Stages of Change, Healthier eating behavior; Test type: Superiority; p = 0.5669, Regression, Logistic; Odds Ratio (OR) = 1.216, 95% CI 2-sided [0.622 to 2.376]
Statistical Analysis 5: Comparison: Health Coaching vs Non-Health Coaching; Stages of Change, Stress behavior; Test type: Superiority; p = 0.1210, Regression, Logistic; Odds Ratio (OR) = 0.622, 95% CI 2-sided [0.341 to 1.134]
Statistical Analysis 6: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Weight reduction; Test type: Superiority; p = 0.8355, Regression, Logistic; Odds Ratio (OR) = 0.928, 95% CI 2-sided [0.461 to 1.872]
Statistical Analysis 7: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Exercise behavior; Test type: Superiority; p = 0.0459, Regression, Logistic; Odds Ratio (OR) = 1.830, 95% CI 2-sided [1.011 to 3.311]
Statistical Analysis 8: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Smoking behavior; Test type: Superiority; p = 0.4650, Regression, Logistic; Odds Ratio (OR) = 0.563, 95% CI 2-sided [0.121 to 2.629]
Statistical Analysis 9: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Healthier eating behavior; Test type: Superiority; p = 0.8303, Regression, Logistic; Odds Ratio (OR) = 0.930, 95% CI 2-sided [0.478 to 1.808]
Statistical Analysis 10: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Stress behavior; Test type: Superiority; p = 0.3254, Regression, Logistic; Odds Ratio (OR) = 1.347, 95% CI 2-sided [0.744 to 2.439]

23. Secondary Outcome: Depression, as Measured by the Beck Depression Inventory (BDI)
Description: The Beck Depression Inventory is a 21-item measure that assesses self-reported symptoms of depression. It has been heavily used in research linking depression to heart disease. Scores range from 0-63, with 0 = minimal depression and 63 = severe depression.
Time Frame: 6 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
units on a scale | 3.85 (0.37) | 5.1 (0.37) | 4.52 (0.37) | 4.43 (0.38)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.0174, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.8694, Regression, Linear

24. Secondary Outcome: Unmanaged Stress as Measured by the Perceived Stress Scale (PSS)
Description: The PSS is a 10 item survey assessing feelings and thoughts of stress. Scores range from 0-40 with higher scores indicating higher perceived stress.
Time Frame: 6 months
Population: Randomization Arms/Groups were regrouped as pre-specified in the study protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 71 | 77 | 69
units on a scale | 10.86 (0.56) | 11.43 (0.56) | 11.07 (0.55) | 11.22 (0.56)
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.4768, Regression, Linear
Statistical Analysis 2: Comparison: Genetic Risk Counseling vs Non-Genetic Risk Counseling; Test type: Superiority; p = 0.8452, Regression, Linear

25. Secondary Outcome: Social Isolation
Description: Single item to assess for availability of support person, where No=no support person.
Time Frame: 6 months
Population: Data is reported for participants who had data available at the 6 month visit. Randomization Arms/Groups were regrouped as pre-specified in the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Coaching | Non-Health Coaching | Genetic Risk Counseling | Non-Genetic Risk Counseling
Number analyzed (Participants) | 75 | 76 | 77 | 74
Participants
  Social Support=No | 3 | 7 | 8 | 2
  Social Support=Yes | 72 | 69 | 69 | 72
Statistical Analysis 1: Comparison: Health Coaching vs Non-Health Coaching; Test type: Superiority; p = 0.5589, Regression, Logistic; Odds Ratio (OR) = 1.591, 95% CI 2-sided [0.335 to 7.544]

ADVERSE EVENTS:
Time Frame: date of consent to 12 months
Arm/Group | Standard Risk Assessment (SRA) | SRA Plus Health Coaching (HC) | SRA Plus Genetic Risk Counseling (GRC) | SRA+HC+GRC
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49 | 0/49 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/49 | 0/49 | 0/52
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49 | 0/49 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Risk Assessment (SRA) (N=50) | SRA Plus Health Coaching (HC) (N=49) | SRA Plus Genetic Risk Counseling (GRC) (N=49) | SRA+HC+GRC (N=52)
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT01884545/Prot_SAP_000.pdf